CLINICAL TRIAL: NCT02126085
Title: Sedation vs. Intubation for Endovascular Stroke TreAtment
Acronym: SIESTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. Silvia Schönenberger, MD, Leading sub-investigator, Principal Investigator: PD Dr. Julian Bösel, MD, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIESTA
Record Dates: First submitted 2014-04-23; First posted 2014-04-29 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Acute Ischemic Stroke
Keywords: ischemic stroke; recanalisation; sedation
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intubation (Active Comparator): Intubation and invasive mechanical ventilation + endovascular recanalisation
  Interventions: Procedure: Endovascular recanalisation
- No Intubation (Experimental): Conscious sedation and non-invasive ventilatory support + endovascular recanalisation
  Interventions: Procedure: Endovascular recanalisation

INTERVENTIONS:
Procedure: Endovascular recanalisation — Endovascular recanalisation by mechanical thrombectomy with e.g. stent retriever device, possibly following intravenous thrombolysis within a "bridging concept"

SUMMARY:
Sedation vs Intubation for Endovascular Stroke TreAtment Trial (SIESTA) is a prospective, randomised controlled, monocentric, two-armed, comparative trial. Patients are randomized 1 : 1 to either non-intubated state or to intubated state for endovascular stroke treatment. Otherwise, no principal differences in intensive care treatment are intended, and standard operating procedures are applied to ensure uniform management decisions in fields such as ventilation, sedation, cardio-vascular and cerebral monitoring and management.

DETAILED DESCRIPTION:
Early recanalization is an important, if not the most important, factor concerning reconstitution of patients´ health in ischaemic stroke. This is the reason why patients with extended stroke are increasingly subjected to an endovascular stroke therapy (EST).

Matter of ongoing debate is how to sedate these patients during intervention. Some clinicians prefer an intubation due to a reduction of patients´movements and therefore potentially lowering complication rates (injury by catheter, aspiration e.g.).

On the other hand retrospective investigations hypothesize that general anaesthesia is associated with peri-interventional hypotension followed by poorer clinical outcome.

The best anaesthaesiologic management in endovascular stroke therapy to this point of time is not known. The investigators therefore designed this study comparing intubated state with general anaesthesia vs. non-intubated state with conscious sedation during EST, focusing on patients´ outcome.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* acute stroke in anterior circulation
* occlusion of carotid artery and/ or middle cerebral artery
* planned mechanical recanalisation
* informed consent from patient or legal representative

Exclusion Criteria:

* age < 18 years
* informed consent not obtainable
* coma
* agitation
* vomiting
* difficult airway management
* additional cerebral hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) after 24 hours | 24 hours
  Neurological improvement of NIHSS 24 hours after intervention

SECONDARY OUTCOMES:
Outcome after 3 month using the modified Rankin Scale (mRS) | 3 month
  Assessing the neurological outcome after 3 months with the mRS.
Inpatient-mortality | Mortality-rate until timepoint of discharge, an expected average of 3 weeks.
Mortality-rate within the first 3 months after intervention. | First 3 months after intervention

OTHER OUTCOMES:
Duration of hospital stay | Participants will be followed until timepoint of discharge, an expected average of 3 weeks.
Periinterventional complications | Evaluation of Adverse Events as a Measure of Safety and Tolerability until timepoint of discharge, an expected average of 3 weeks.
Achieved recanalisation grade | Duration of intervention with an expected average of 2 hours
  Recanalisation status is classified according to the Thrombolysis in Cerebral Infarction classification (TICI).

CONTACTS AND LOCATIONS:
Overall Officials: Julian Bösel, PD, Principal Investigator — Department of Neurology, University Hospital Heidelberg
Locations (1):
- Department of Neurology, University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Lees KR, Bluhmki E, von Kummer R, Brott TG, Toni D, Grotta JC, Albers GW, Kaste M, Marler JR, Hamilton SA, Tilley BC, Davis SM, Donnan GA, Hacke W; ECASS, ATLANTIS, NINDS and EPITHET rt-PA Study Group; Allen K, Mau J, Meier D, del Zoppo G, De Silva DA, Butcher KS, Parsons MW, Barber PA, Levi C, Bladin C, Byrnes G. Time to treatment with intravenous alteplase and outcome in stroke: an updated pooled analysis of ECASS, ATLANTIS, NINDS, and EPITHET trials. Lancet. 2010 May 15;375(9727):1695-703. doi: 10.1016/S0140-6736(10)60491-6. PMID 20472172
- [Background] Rha JH, Saver JL. The impact of recanalization on ischemic stroke outcome: a meta-analysis. Stroke. 2007 Mar;38(3):967-73. doi: 10.1161/01.STR.0000258112.14918.24. Epub 2007 Feb 1. PMID 17272772
- [Background] Nogueira RG, Liebeskind DS, Sung G, Duckwiler G, Smith WS; MERCI; Multi MERCI Writing Committee. Predictors of good clinical outcomes, mortality, and successful revascularization in patients with acute ischemic stroke undergoing thrombectomy: pooled analysis of the Mechanical Embolus Removal in Cerebral Ischemia (MERCI) and Multi MERCI Trials. Stroke. 2009 Dec;40(12):3777-83. doi: 10.1161/STROKEAHA.109.561431. Epub 2009 Oct 29. PMID 19875740
- [Background] Bosel J, Hacke W, Bendszus M, Rohde S. Treatment of acute ischemic stroke with clot retrieval devices. Curr Treat Options Cardiovasc Med. 2012 Jun;14(3):260-72. doi: 10.1007/s11936-012-0172-y. PMID 22392611
- [Background] McDonagh DL, Olson DM, Kalia JS, Gupta R, Abou-Chebl A, Zaidat OO. Anesthesia and Sedation Practices Among Neurointerventionalists during Acute Ischemic Stroke Endovascular Therapy. Front Neurol. 2010 Nov 11;1:118. doi: 10.3389/fneur.2010.00118. eCollection 2010. PMID 21188256
- [Background] Davis MJ, Menon BK, Baghirzada LB, Campos-Herrera CR, Goyal M, Hill MD, Archer DP; Calgary Stroke Program. Anesthetic management and outcome in patients during endovascular therapy for acute stroke. Anesthesiology. 2012 Feb;116(2):396-405. doi: 10.1097/ALN.0b013e318242a5d2. PMID 22222475
- [Derived] Tosello R, Riera R, Tosello G, Clezar CN, Amorim JE, Vasconcelos V, Joao BB, Flumignan RL. Type of anaesthesia for acute ischaemic stroke endovascular treatment. Cochrane Database Syst Rev. 2022 Jul 20;7(7):CD013690. doi: 10.1002/14651858.CD013690.pub2. PMID 35857365
- [Derived] Schonenberger S, Uhlmann L, Ungerer M, Pfaff J, Nagel S, Klose C, Bendszus M, Wick W, Ringleb PA, Kieser M, Mohlenbruch MA, Bosel J. Association of Blood Pressure With Short- and Long-Term Functional Outcome After Stroke Thrombectomy: Post Hoc Analysis of the SIESTA Trial. Stroke. 2018 Jun;49(6):1451-1456. doi: 10.1161/STROKEAHA.117.019709. Epub 2018 May 2. PMID 29720440
- [Derived] Schonenberger S, Uhlmann L, Hacke W, Schieber S, Mundiyanapurath S, Purrucker JC, Nagel S, Klose C, Pfaff J, Bendszus M, Ringleb PA, Kieser M, Mohlenbruch MA, Bosel J. Effect of Conscious Sedation vs General Anesthesia on Early Neurological Improvement Among Patients With Ischemic Stroke Undergoing Endovascular Thrombectomy: A Randomized Clinical Trial. JAMA. 2016 Nov 15;316(19):1986-1996. doi: 10.1001/jama.2016.16623. PMID 27785516